CLINICAL TRIAL: NCT06045169
Title: The Effects of Muscle Energy Techniques on Pain and Quality of Life in Young Females With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/15
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Quasi Experimental Pre-test Post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Other): Post isometric relaxation with participants using 20% of their maximum voluntary contraction will be given to global muscles of core commonly involved in primary dysmenorrhea glutus maximus, Illiopsoas and pirifirmis. Post isometric contraction will be held for 6 to 10 seconds followed by 15 o 30 seconds stretch, rst time will be 5 seconds in between repetations and number of repetations will be 3-5.
  Interventions: Procedure: Post Isometric Relaxation

INTERVENTIONS:
Procedure: Post Isometric Relaxation — Post isometric relaxation with participants using 20% of their maximum voluntary contraction will be given to global muscles of core commonly involved in primary dysmenorrhea glutus maximus, Illiopsoas and pirifirmis. Post isometric contraction will be held for 6 to 10 seconds followed by 15 o 30 seconds stretch, rst time will be 5 seconds in between repetations and number of repetations will be 3-5.

SUMMARY:
This study will be a quasi experimental study in which females aged 18 - 30 years with primary dysmenorrhea will be recruited in single group. They will be given a total of 3 sessions of treatment during a period of one menstrual cycle (One Week). Before and after the introduction of intervention pain and quality of life of participants will be assessed.

DETAILED DESCRIPTION:
Primary Dysmenorrhea is one of the most prevalent gynecological conditions which impacts the quality of life of young females.Primary dysmenorrhea is defined as cramping like pain during menstruation cycle without the presence of any pelvic pathology it is associated with symptoms like headache,vomitting and irritability.The aim of our study is to determine the effects of muscle energy technique in young females with primary dysmenorrhea in terms of pain and quality of life.This study will be a Quasi Experimental study.It will be conducted at Foundation university college of physical therapy.Paticipants will complete WALIDD scale,NPRS and WHOQOL at baseline and then after intervention.All participants will receive post isometric relaxation of global muscles of core commonly involved in primary dysmenorrhea(Gluteus Maximus,Illiopsoas and Piriformis).Post isometric relaxation technique will be applied to all the participants with participants using 20% of their maximum voluntary contractio with held time of 6-10 seconds followed by 15 to 30 seconds stretch,rest time of 5 seconds between each repetitions and 3-5 repetions.There will be a total of 3 sessiond of treatment(1st on second day of menstruation,2nd on fourth day of menstruatio and 3rd on seventh day of menstruation)during a period of one week (one menstraul cycle).

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 - 30
* Primary Dysmenorrhea
* Unmarried

Exclusion Criteria:

* Not on any contraceptive medicine for treatment of pelvic pathology
* Secondary Dysmenorrhea and other issues such as endometriosis, Pelvic inflammatory disease, Ovarian cyst

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female between ages 18-30 years
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 week
  Pain will be measured using numeric pain rating scale which is an 10 point scale scored from zero indicating no pain and 10 indicating worst pain.

SECONDARY OUTCOMES:
Quality of life of participant | 1 week
  Quality of life will be measured by WHOQOL-bref (World Health questionnaire for quality of life) which is valid and reliable tool for measuring quality of life with 26 instruments, Each individual item score from one to five on response scale.
WALIDD | 1 week
  Working ability, Location, Intensity, Days of pain, Dysmenorrhea (WALIDD) is a scale with four categories Score of each category is added to find out the total level of severity of dysmenorrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan